CLINICAL TRIAL: NCT00770432
Title: A Randomized, Placebo-Controlled, Double-Blind, Trial of Polyethylene Glycol 3350 Laxative for the Treatment of Occasional Constipation.
Brief Title: Study Comparing PEG 3350 Laxative to Placebo in the Treatment of Occasional Constipation (Study CL2007-12)(P08216)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18130; CL2007-12; P08216 (Other: Merck)
Record Dates: First submitted 2008-10-09; First posted 2008-10-10 (Estimated); Results first posted 2009-08-12 (Estimated); Last update posted 2018-10-02 (Actual); Status verified 2018-09

CONDITIONS: Constipation
Keywords: Human Experimentation
MeSH Terms: conditions — Constipation | interventions — polyethylene glycol 3350; Solutions

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Polyethylene glycol 3350 powder for solution (Active Comparator): MiraLAX® (polyethylene glycol 3350 powder for solution)
  Interventions: Drug: Polyethylene glycol 3350
- Placebo (Placebo Comparator): MALTRIN 500® M500 (maltodextrin 500)
  Interventions: Other: Placebo, maltodextrin 500 powder for solution

INTERVENTIONS:
Drug: Polyethylene glycol 3350 — Polyethylene glycol 3350 powder for solution. Single dose (17 grams in 4 to 8 ounces of beverage) for 7 days.
  Other Names: MiraLAX®
  Arms: Polyethylene glycol 3350 powder for solution
Other: Placebo, maltodextrin 500 powder for solution — Maltodextrin 500 powder for solution, One single dose (one capful) in any 4 - 8 ounces beverage for 7 days.
  Other Names: MALTRIN® 500 powder for solution
  Arms: Placebo

SUMMARY:
Randomized, placebo-controlled, double blind study. 203 subjects entered the study to compare the effect on occasional constipation of polyethylene glycol 3350 to placebo. Subjects took one of study treatments up to 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Subjects (or parents/guardians of minors) must demonstrate their willingness to participate (or to have their children/wards participate) in the study and comply with its procedures by signing a written informed consent. Minor subjects must provide written assent.
* Subjects must be 17 years of age or older.
* Subjects must present with a current diagnosis of untreated constipation for 7 days or less based on having signs/symptoms of straining and hard or lumpy stools OR the inability to have a BM within 48 hours prior to randomization into the trial.
* Subjects must be OTC laxative users for the treatment of occasional constipation (defined as using a nonprescription laxative to treat at least 3 episodes of constipation within the last 12 months prior to randomization).
* Subjects must be willing to use study drug for up to 7 days as directed, and must agree to record bowel movement (frequency, consistency, etc.) accurately and consistently in a daily diary, and make two clinic visits.
* Subjects must be otherwise in good health, as determined by physical exam and medical history.
* Subjects must agree not to use any other products to treat their constipation during the course of the study.
* Subjects must agree not to use any medication known to cause constipation during the course of the study.
* Subjects must agree to maintain a similar diet from the week prior to randomization through end of study.
* Female subjects must be either surgically sterile, 2 years post-menopausal, or they attest that they are using an acceptable method of contraception (including hormonal birth control, IUD, double barrier methods, or vasectomized partner). In females of childbearing potential, the urine pregnancy test (HCG) must be negative at Baseline.
* Subjects must be able to read the diaries in English.

Exclusion Criteria:

* Subjects currently under a doctor's care and treatment for constipation.
* Subjects having current constipation episode for more than one week prior to randomization.
* Subjects that have a history of chronic constipation due to any underlying cause (inflammatory bowel disease, etc.).
* Subjects have a history of more than 3 months of constipation in the past year.
* Subjects have severe abdominal pain as the predominant constipation symptom.
* Subjects who have previously used a polyethylene glycol laxative.
* Subjects who have celiac disease or known gluten sensitivity.
* Subjects who have a history of colorectal cancer, anal abscess, anal fistula, anal fissure, anal stenosis, gastric retention or obstruction, bowel resection, rectocele, or colostomy.
* Subjects with known renal or hepatic insufficiency.
* Subjects with gastrointestinal bleeding or acute infection.
* Subjects with a history of alcohol or drug abuse.
* Subjects with a history of psychiatric disorders.
* Subjects with a history of significant ongoing medical problems, including kidney disease, or who are scheduled for surgical procedures.
* Subjects currently taking or taken within 7 days of randomization a concomitant medication that causes constipation including for example opiates, antidepressants, SSRI's, antimotility agents, and anticholinergics, etc.
* Subjects who plan to use laxatives during the treatment period other than the study medication.
* Subjects who, in the opinion of the investigator, should not be included in the study for any reason, including inability to follow study procedures.
* Subjects who have participated in an investigational clinical surgical, drug or device study within the past 30 days.
* Subjects who are pregnant or lactating.
* Subjects who are allergic to polyethylene glycol or maltodextrin.
* Subjects who are employed or have immediate family members employed by a company that manufactures laxative products.

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2007-11; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

REFERENCES:
- [Derived] McGraw T. Polyethylene glycol 3350 in occasional constipation: A one-week, randomized, placebo-controlled, double-blind trial. World J Gastrointest Pharmacol Ther. 2016 May 6;7(2):274-82. doi: 10.4292/wjgpt.v7.i2.274. PMID 27158544

RESULTS

PARTICIPANT FLOW:
Groups:
- Polyethylene Glycol 3350 Powder for Solution: MiraLAX® (polyethylene glycol 3350 powder for solution). Single dose (17 grams dissolved in 4 to 8 ounces of beverage) for 7 days.
- Placebo: MALTRIN 500® M500 (maltodextrin 500 powder for solution). Single dose (one capful) in 4 to 8 ounces of beverage for 7 days.
Period: Overall Study
Arm/Group | Polyethylene Glycol 3350 Powder for Solution | Placebo
Started | 102 | 101
Completed | 98 | 94
Not Completed | 4 | 7
Not completed — Other | 4 | 6
Not completed — Non-compliance | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Polyethylene Glycol 3350 Powder for Solution | Placebo | Total
Number analyzed (Participants) | 102 | 101 | 203
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.8 (12.52) | 45.0 (14.15) | 45.4 (13.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 68 | 145
  Male | 25 | 33 | 58

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Complete Resolution at the Final Visit
Description: A resolution was recorded if the participant has no occurrence of two or more consecutive unsuccessful bowel movements for the rest of the study following the first successful bowel movement.
Time Frame: 24 hours to 3 days after last dose of seven day treatment period.
Population: Per-Protocol Population
Measure: Number; unit: Participants
Arm/Group | Polyethylene Glycol 3350 Powder for Solution | Placebo
Number analyzed (Participants) | 98 | 94
Participants | 36 | 23
Statistical Analysis 1: Comparison: Polyethylene Glycol 3350 Powder for Solution vs Placebo; Test type: Superiority or Other; p = 0.0595, Cochran-Mantel-Haenszel; The Cochran-Mantel-Haenszel adjusted for study site (the smallest study sites were pooled according to a pre-specified rule)

ADVERSE EVENTS:
Arm/Group | Polyethylene Glycol 3350 Powder for Solution | Placebo
Serious Adverse Events (participants affected / at risk) | 0/102 | 0/101
Other Adverse Events (participants affected / at risk) | 11/102 | 11/101
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Polyethylene Glycol 3350 Powder for Solution (N=102) | Placebo (N=101)
Headache (Nervous system disorders) | 11 (14) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other